CLINICAL TRIAL: NCT06904404
Title: Physiologic Phacofluidics: Ghost Protocol
Status: Completed | Type: Observational
Sponsor: Wolfe Eye Clinic (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Edward Hsu Hu, Primary Investigator, Wolfe Eye Clinic
Other Study IDs: 83557125
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Cataract
Keywords: phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High IOP setting: Traditional High (65mm Hg) IOP phacoemulsification settings
  Interventions: Procedure: Cataract surgery at high IOP
- Low IOP Setting: Physiologic Low (20 mm Hg) IOP phacoemulsification settings
  Interventions: Procedure: Cataract surgery at low IOP

INTERVENTIONS:
Procedure: Cataract surgery at high IOP — Cataract surgery at high IOP (conventional)
  Groups: High IOP setting
Procedure: Cataract surgery at low IOP — Cataract surgery at low IOP
  Groups: Low IOP Setting

SUMMARY:
The goal of this clinical trial is to investigate the early post-operative benefits of performing phacoemulsification at physiologic intraocular pressures. The main questions it aims to answer are:

* Is there less post operative corneal edema?
* Is there less post operative inflammation?
* Is the post operative vision better? Participants will undergo phacoemulsification cataract surgery with either high or low IOP settings Researchers will compare post op corneal edema, inflammatory marker levels and vision

DETAILED DESCRIPTION:
Methods:

Study population Inclusion Criteria

* Patients without prior ocular surgery both eyes
* Adult patients with visually significant cataract with WHO-World Health Organization NUC grade 2-3
* First eye only undergoing uncomplicated cataract surgery
* Unremarkable systemic history; controlled diabetes with HbA1c <7%
* Unremarkable ocular health
* Anterior chamber depth ACD >2.04mm10
* Age range 55-95

Exclusion Criteria:

* Prior ocular surgery including corneal refractive surgery, cataract surgery in fellow eye
* Thin corneas (<490 microns)
* Complicated (use of pupil expansion devices) or prolonged cataract surgeries (>15 mins) with post-operative complications (IOP spike >30mmHg), severe punctate keratitis

Approximately 66 patients will be identified and included in the study. Patients at the day of surgery sign up will be randomized to high (65mmHg) vs low IOP (20mmHg) using a random online number generator; Even will be high IOP; Odd will be low IOP. Patients will undergo standard cataract surgery with equivalent vacuum and aspiration rates in both groups for the duration of the entire cataract surgery; IOP settings will be set at high vs low IOP but may be adjusted if necessary for the safety of the patient.

In all procedures, the intraocular lens (IOL) implanted and the ophthalmic viscosurgical device (OVD) materials used will be standardized to the same materials and are part of routine surgery. Cumulative dissipated energy (CDE) and surgical duration will be collected for all patients. An intraoperative aqueous sample 100-150µL will be collected at the end of the case 2 minutes after OVD removal and immediately transferred on dry ice to a laboratory, stored at -80°C until analysis as established in prior protocol. The extraction of aqueous sample will not require additional incisions.

All subjects will be prescribed the standard post-operative cataract surgery medications (not specific to study). Post-operative visits by the masked sub-investigator will perform the following procedures at 4hrs (early post-op), POD#1 (20-24hrs), POW#1:

Post-op Procedures Baseline Visit1 (4hrs) Visit2 (20-24hrs) Visit3 (1 week) Pachymetry X X X X Visual acuity BCVA UCVA/PHVA UCVA/PHVA UCVA/PHVA Slit Lamp- Cell /Flare X X X X

Pachymetry: a painless, simple test where a probe is gently placed on the front of the eye to measure the thickness of the cornea.

Best-corrected visual acuity (BCVA): this test is used to determine the smallest letters that can be read on a standardized chart. Un-corrected visual acuity (UCVA): the smallest letter that can be read unaided. Pinhole visual acuity (PHVA): the smallest letter that can be read without the interference of optical problems.

Slit lamp exam: a microscope is used to provide a magnified view of different parts of the eye and to determine inflammation (cell/flare) that is common with any ophthalmic surgery.

Visual acuity and slit lamp examinations are part of routine post-operative care.

Pachymetry measurements are for research purposes to determine if there's less corneal swelling after cataract surgery in the lower IOP group.

The primary end point is: difference in CCT post-op at 4 hours between High vs Low IOP groups.

Secondary endpoints include: CCT at POD#1 and POW#1, Cell/Flare at POHr4 and POD1, and inflammatory markers: levels of prostaglandin IL-6, IL-8, IL-Iβ, TNF-α, PGE2, MCP-1. Aqueous samples will be sent with de-identified patient information and aqueous analysis will be performed by the University of California, Irvine Molecular Biology and Biochemistry Labs. The laboratory will be masked to which treatment the subject received and will only provide the aqueous analysis report for the study.

Any adverse events (AE) will be recorded in subject's medical charts as well as an adverse event log. AEs are classified as serious or non-serious; expected or unexpected; and study-related, possibly study-related, or not study-related. Serious AEs will be reported immediately to the regulatory authorities as per standard of care. The potential risks involved are that of standard cataract surgery with potential complications and side effects associated with any surgical procedure. These include but are not limited to: infection, macular edema, increased IOP, general risk of anesthesia and surgery, bleeding in the eye, and decreased vision. Some potential benefits include: improved visual acuity, decreased glare symptoms, lowered IOP, and faster visual recovery.

Analysis:

Primary endpoint: Difference in mean CCT change at 4 hrs post-surgery between high vs low IOP will be assessed using t-test with a P-value <0.05. Descriptive statistics will be used for the other secondary endpoints

Sample Size Justification:

The expected mean CCT change between the high vs low groups is hypothesized to be 32um, with a standard deviation of 40um. With a Type I/II error rate of alpha=0.05 and power=0.85, a sample size of 56 eyes are needed; additional 10 eyes to account for ~15 attrition; N=66

Data Collection and Management:

Data is recorded in a manner that reduces the risk of a breach of confidentiality. Password protected Microsoft Excel files will be utilized for this study and only accessible by authorized study personnel.

Ethical and Regulatory Considerations:

The study is conducted in accordance with the following:

Protocol and study-related plans and documents

* Local regulations, as applicable
* Good Clinical Practices, as outlined in the ICH Harmonized Tripartite Guideline for GCP (ICH

E6(R2))Ethical and Regulatory Considerations:

The study is conducted in accordance with the following:

* Protocol and study-related plans and documents
* Local regulations, as applicable
* Good Clinical Practices, as outlined in the ICH Harmonized Tripartite Guideline for CP (ICH E6(R2))
* The ethical principles established by the Declaration of Helsinki
* Regional participant data protection laws and regulations
* Local IRB requirements

Institutional Review Board (IRB):

The study site will maintain an accurate and complete record of all reports, documents and other submissions made to the Institutional Review Board (IRB) concerning this protocol.

The investigator must supply ongoing study progress reports to the IRB, per local requirements, protocol deviations and amendments. In addition, the investigator must notify the IRB at the closure of the study.

Informed Consent:

It is the responsibility of the investigator and clinical coordinator to inform each subject of the purpose of this study, including possible risks and benefits and document the informed consent process in the subject's chart. Prior to entry into the study or initiation of any study-related testing, the subject must read, sign and date the informed consent form. If the subject's vision is impaired to the point where they cannot read the informed consent document, the document will be read to the subject. The person executing the consent must also sign and date the consent form. One original informed consent form is to be retained by the study site and a copy is to be given to the subject.

Protocol Amendments:

This protocol must be followed as written. Any change or addition to this protocol that impacts subject safety, or the validity of the study requires a written protocol amendment that must be approved in writing by the IRB and any required regulatory authorities before implementation.

Record Keeping and Retention:

Data generated for the study should be stored in a limited-access file area and be accessible only to study personnel of the site. All reports and communications relating to study participants will identify participants only by subject identification number. Complete subject identification will be kept by the investigator. This information will be treated with strict adherence to professional standards of confidentiality.

The Investigator will retain a copy in the study file:

* A copy of the IRB approved informed consent form
* All original informed consent forms with required signatures
* All participant source documents, etc.
* All IRB correspondence (i.e., informed consent [including any approved revisions], protocol, AE, advertisements, newsletters).

Confidentiality:

All clinical study findings and documents are regarded as confidential. Study documents (protocols and other material) must be stored appropriately to ensure their confidentiality.

The anonymity of participants must be maintained per applicable local and national laws. Subjects are specified on all documents by subject number but not by name. Documents that identify the subject, e.g., the signed ICF, must be maintained in confidence by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients without prior ocular surgery both eyes
* Adult patients with visually significant cataract with WHO-World Health Organization NUC grade 2-3
* First eye only undergoing uncomplicated cataract surgery
* Unremarkable systemic history; controlled diabetes with HbA1c <7%
* Unremarkable ocular health
* Anterior chamber depth ACD >2.04mm10
* Age range 55-95

Exclusion Criteria:

* Prior ocular surgery including corneal refractive surgery, cataract surgery in fellow eye
* Thin corneas (<490 microns)
* Complicated (use of pupil expansion devices) or prolonged cataract surgeries (>15 mins) with post-operative complications (IOP spike >30mmHg), severe punctate keratitis

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visually significant cataract patients with no prior history of cataract surgery
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward H Hu, MD PhD, Principal Investigator — Wolfe Eye Clinic
Locations (1):
- Wolfe Eye Clinic Cedar Rapids (Hiawatha), Hiawatha, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cyril D, Brahmani P, Prasad S, Rashme VL, R S, Kamble NR, Balakrishnan L, Nagu K, Shekhar M. Comparison of two phacoemulsification system handpieces: prospective randomized comparative study. J Cataract Refract Surg. 2022 Mar 1;48(3):328-333. doi: 10.1097/j.jcrs.0000000000000769. PMID 34371511
- [Background] Vasavada AR, Praveen MR, Vasavada VA, Vasavada VA, Raj SM, Asnani PK, Garg VS. Impact of high and low aspiration parameters on postoperative outcomes of phacoemulsification: randomized clinical trial. J Cataract Refract Surg. 2010 Apr;36(4):588-93. doi: 10.1016/j.jcrs.2009.11.009. PMID 20362850
- [Background] Lundberg B, Jonsson M, Behndig A. Postoperative corneal swelling correlates strongly to corneal endothelial cell loss after phacoemulsification cataract surgery. Am J Ophthalmol. 2005 Jun;139(6):1035-41. doi: 10.1016/j.ajo.2004.12.080. PMID 15953433
- [Background] Suzuki H, Igarashi T, Takahashi H. Effect of a new phacoemulsification and aspiration handpiece on anterior chamber stability. J Cataract Refract Surg. 2023 Jan 1;49(1):91-96. doi: 10.1097/j.jcrs.0000000000001071. PMID 36201661
- [Background] Kaup S, Pandey SK. Cataract surgery in patients with Fuchs' endothelial corneal dystrophy. Community Eye Health. 2019;31(104):86-87. No abstract available. PMID 31086438
- [Background] Liu YC, Setiawan M, Ang M, Yam GHF, Mehta JS. Changes in aqueous oxidative stress, prostaglandins, and cytokines: Comparisons of low-energy femtosecond laser-assisted cataract surgery versus conventional phacoemulsification. J Cataract Refract Surg. 2019 Feb;45(2):196-203. doi: 10.1016/j.jcrs.2018.09.022. Epub 2018 Dec 6. PMID 30528516
- [Background] De Maria M, Iannetta D, Cimino L, Coassin M, Fontana L. Measuring Anterior Chamber Inflammation After Cataract Surgery: A Review of the Literature Focusing on the Correlation with Cystoid Macular Edema. Clin Ophthalmol. 2020 Jan 9;14:41-52. doi: 10.2147/OPTH.S237405. eCollection 2020. PMID 32021067
- [Background] Schultz T, Joachim SC, Kuehn M, Dick HB. Changes in prostaglandin levels in patients undergoing femtosecond laser-assisted cataract surgery. J Refract Surg. 2013 Nov;29(11):742-7. doi: 10.3928/1081597X-20131021-03. PMID 24203805
- [Background] Feng MT, Belin MW, Ambrosio R Jr, Grewal SP, Yan W, Shaheen MS, McGhee C, Maeda N, Neuhann TH, Burkhard Dick H, Alageel SA, Steinmueller A. Anterior chamber depth in normal subjects by rotating scheimpflug imaging. Saudi J Ophthalmol. 2011 Jul;25(3):255-9. doi: 10.1016/j.sjopt.2011.04.005. Epub 2011 Apr 30. PMID 23960933

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the recruitment period, 66 subjects were enrolled. One subject, the surgeon deviated from the intra-operative study protocol due to the density of the lens by using additional instrumentation (miLoop) to remove the lens. One subject had CCT performed on the wrong eye, one subject missed their 1-week follow-up visit. Two subjects had CCT readings performed with a Pentacam as opposed to a Lenstar (instrument malfunction).
Units Other Than Participants: eyes
Groups:
- Low IOP: N= 30
- High IOP: N=31
Period: Overall Study
Arm/Group | Low IOP | High IOP
Started | 33; 66 eyes | 33; 66 eyes
Completed | 30; 60 eyes | 31; 62 eyes
Not Completed | 3; 6 eyes | 2; 4 eyes

BASELINE CHARACTERISTICS:
Groups:
- Low IOP: Patients randomized to low (20 mmHg) IOP surgical settings using the Active Sentry handpiece
- High IOP: Patients randomized to High (65 mmHg) IOP surgical settings using the Active Sentry handpiece
- Total: Total of all reporting groups
Arm/Group | Low IOP | High IOP | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (1.1) | 70.5 (0.8) | 70.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Early Post Operative Central Corneal Thickness
Description: 4 hours post operatively central corneal thickness assessment
Time Frame: 4 hours post operatively
Population: Those that completed all follow-ups
Measure: Mean (Standard Deviation); unit: microns
Groups:
- High IOP Group; Low IOP Group: Patients randomized to either high (65 mmHg) or low (20 mmHg) IOP surgical settings using the Active Sentry handpiece.
Arm/Group | High IOP Group | Low IOP Group
Number analyzed (Participants) | 31 | 30
microns | 623.9 (9.9) | 650.2 (11.9)

2. Secondary Outcome: IL-IB From Aqueous Sample
Description: Early post op aqueous inflammatory marker of IL-IB level assessment
Time Frame: 2 minutes after cataract surgery completion
Population: Those completed surgery & follow-ups
Measure: Mean (Standard Deviation); unit: pg/ML
Groups:
- Low IOP; High IOP: Patients randomized to either high (65 mmHg) or low (20 mmHg) IOP surgical settings using the Active Sentry handpiece.
Arm/Group | Low IOP | High IOP
Number analyzed (Participants) | 30 | 31
pg/ML | 0.6130 (0.0911) | 0.6806 (0.0935)

ADVERSE EVENTS:
Time Frame: 6 month
Description: Adverse events were monitored/assessed but no patients had any adverse events in the study
Groups:
- Low IOP Group; High IOP Group: No adverse events, product issues, or other safety events were observed in this study.
Arm/Group | Low IOP Group | High IOP Group
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT06904404/Prot_SAP_001.pdf